CLINICAL TRIAL: NCT01910168
Title: A Single Center Study to Collect Samples From SMA Patients for Biomarker Analysis
Brief Title: A Study to Collect Blood Samples From Patients With Spinal Muscular Atrophy for Biomarker Analysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: BE29002
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
In this single center study blood samples for biomarker analysis will be collected from patients with spinal muscular atrophy. Up to 21 mL blood will be drawn from eligible patients at a single visit.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as 5q-autosomal recessive spinal muscular atrophy (SMA) type I, II or III as judged by their neurologist upon diagnosis
* Ability and willingness to provide blood samples
* Willingness (by the patient or patient's parents or legal guardian) to complete to their best ability a questionnaire which requests specific clinical and genetic information
* Able to participate and willing to give written informed consent or assent. Informed consent will be obtained from the patient, or the patient's parent or legal guardian.

Exclusion Criteria:

* Any known genetic condition other than spinal muscular atrophy, unless it is not interfering with the purpose of this study based on the Sponsor's judgment
* Participation in a clinical trial (except observational studies) within the previous 14 days
* Donation of blood or significant blood loss within three months prior to screening
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of this study, or that would, in the opinion of the investigator, pose an unacceptable risk to the patient in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with spinal muscular atrophy
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
SMN1/SMN2 detection in blood by mRNA assay | 1 day

SECONDARY OUTCOMES:
SMN protein level in blood/lymphocytes | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Kalamazoo, Michigan
  - Salt Lake City, Utah